CLINICAL TRIAL: NCT02860533
Title: iPhone App Compared to Standard RR-measurement During Stress Testing
Brief Title: iPhone App Compared to Standard Riva-Rocci (RR)-Measurement During Stress Testing
Acronym: iPARRDeltaBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-00871
Record Dates: First submitted 2016-07-20; First posted 2016-08-09 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Blood Pressure
Keywords: Blood pressure; smartphone App; Hypertension; Stress testing; Prevention; Cardiovascular risk factors
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood pressure measurement (Experimental): six repetitive blood pressure measurements with iPhone and conventional oscillometric cuff device during stress testing will be performed
  Interventions: Device: cuff device; Device: iphone

INTERVENTIONS:
Device: cuff device — Measurement of blood pressure during stress testing with cuff device
Device: iphone — Measurement of blood pressure during stress testing with iPhone

SUMMARY:
The iPARR DELTA BP Study is designed to evaluate whether a new smartphone app using the photoplethysmography signal of the inbuilt camera can measure blood pressure (BP) fluctuations with sufficient correlation compared to the goldstandard oscillometric BP measurements. Investigators will recruit patients who are scheduled for a routine treadmill stress test and assess their blood pressure before and right after the test with the smartphone app and the standard BP measurements on the opposite upper extremity. Pronounced BP fluctuations are encountered during vigorous activities. The primary endpoint of the iPARR DELTA BP Study is the correlation of the absolute difference of subsequent measurements between both techniques. If the relative chances of BP fluctuations are sufficiently assessed with this new device, BP fluctuations could be monitored continuously after calibration.

ELIGIBILITY:
Inclusion Criteria:

- able to give informed consent

Exclusion Criteria:

* atrial fibrillation
* medical reasons why blood pressure measurement is not possible at the upper extremity (Shunt, Lymphedema)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Absolute difference between conventional blood pressure measurements and the corresponding iPhone blood pressure estimations | 1 day
  Difference between the delta of two sequential oscillometric measurements and the delta of the two corresponding blood pressure estimates calculated from the PPG signal of an iPhone 4S

SECONDARY OUTCOMES:
Number of measurement failures | 1 day
  Number of measurements that cannot be analyzed due to bad signal quality of the Photoplethysmography (PPG) signal

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No